CLINICAL TRIAL: NCT06739473
Title: Total-body Glucose Utilization in Obesity
Acronym: TOTAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, professor, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: T335/2022
Record Dates: First submitted 2024-09-29; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Overweight
Keywords: obesity; radiowater; PET
MeSH Terms: conditions — Obesity; Overweight | interventions — Motion Pictures; Cold Temperature

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TOTAL dose test (Experimental): The aim of the studies performed in this arm (8 subjects) is to test the lowest dose of H2[15O]O (radiowater) for the Siemens Quadra PET/CT scanner. Each participant will be studied once with the scanner with 4 different doses (25-700 MBq) of H2[15O]O, each repeated 2 times
  Interventions: Radiation: H2[15O]O PET/CT
- TOTAL (Experimental): The participants in this arm will undergo two PET visits. On one visit the effects of visual stimuli or cold on whole body perfusion will be studied with H2[15O]O PET/CT. On the second visit whole-body insulin sensitivity is studied with [18F]fluorodeoxyglucose PET/CT, and the acute and delayed effects of intravenous insulin on blood flow will be studied with H2[15O]O PET/CT.
  Interventions: Behavioral: Movies; Behavioral: Cold; Drug: Hyperinsulinemic euglycemic clamp; Radiation: H2[15O]O PET/CT; Radiation: [18F]FDG PET/CT; Drug: CEUS or Contrast enhanced Ultrasound

INTERVENTIONS:
Behavioral: Movies — Participants will watch eight short movie clips, and the changes different emotions evoked by the clips will be studied using H2[15O]O PET/CT.
  Arms: TOTAL
Behavioral: Cold — Participants will be studied with H2[15O]O PET/CT while one of their legs will be exposed to cold to study the effects of cold stimulus on whole-body blood flow.
  Arms: TOTAL
Drug: Hyperinsulinemic euglycemic clamp — Participants will be administered intravenous fast acting insulin (NovoRapid, Novo Nordisk, 1 mU/m2 body surface area/min) together with 20 % glucose to maintain normal glucose values (5.0 mmol/L) to study the effects of insulin on whole body blood flow with H2[15O]O PET/CT, and to assess tissue insulin-stimulated glucose uptake with [18F]FDG PET/CT.
  Arms: TOTAL
Radiation: H2[15O]O PET/CT — H2[15O]O PET/CT, with a dose of 25-700 MB/bolus repeated 2-8 times per scan.
Radiation: [18F]FDG PET/CT — Whole-body [18F]FDG PET/CT scan to study tissue glucose uptake, dose 100 MBq
  Arms: TOTAL
Drug: CEUS or Contrast enhanced Ultrasound — Contrast-enhanced ultrasound of left forearm muscles is performed during fasting and after 30-40 minutes of hyperinsulinemia
  Arms: TOTAL

SUMMARY:
There are three goals for this study. One is to investigate how different emotions and exposure to cold affect blood flow in the body. The second aim is to study how insulin affects blood flow and tissue glucose uptake, and to study whether this effect is altered in obesity. Last, the study focuses on establishing the lowest dose of a PET radiotracer, oxygen-15 labelled water, that can be used in clinical studies with a new whole-body PET scanner.

DETAILED DESCRIPTION:
The study consists of two separate parts: the dose escalation study and the part studying the effects of emotions and insulin on blood flow.

All participants will first undergo a screening visit starting with signing an informed consent form. Then they will undergo a physical examination, are interviewed about their medical history. Finally, some routine laboratory tests are collected, and a 75 g oral glucose tolerance test is performed. The participants who are eligibile for the study will continue to the PET studies.

The dose escalation study will be completed first. In this 8 participants will be studied once with Siemens Biovision Quadra PET/CT scanner. They will receive eight doses of oxygen-15 labelledradiowater (H2[15O]O) ranging from 25 to 700 MBq, with each dose repeated twice to evaluate repeatability of each dose. These participants will not undergo any further studies.

For the other subjects, there will be two more PET study visits.

On the first visit, the effects of emotions, evoked by short movie clips or cold exposure of one leg, on whole-body blood flow will studied with oxygen-15 labelled radiowater. Each participant will be studied 8 times in one session, with repeated H2[15O]O boluses of 400 MBq followed by 7.5 min dynamic PET scans with Siemens Biovision Quadra PET/CT scanner and a 5 min recovery and wash-out period.

On the other visit the effects of insulin on circulation will be studied by performing a hyperinsulinemic, euglycemic clamp during the PET scan. During the clamp, fast-acting insulin (NovoRapid, NovoNordisk) is administered intravenously at a fixed rate (40 mU/m2 body surface area/min). Plasma glucose is monitored every 5-10 minutes, and 20 % glucose is administered at a varying rate to maintain euglycemia (5.0 mmol/L).

At the scanner a fasting H2[15O]O PET/CT scan (400 MBq) will be performed first. After this, the hyperinsulinemic, euglycemic clamp is started, and the radiowater scans are repeated 10 minutes and 50 minutes into the insulin infusion. 60 minutes after the start of clamp, 100 MBq of glucose analogue tracer [18F]fluorodeoxyglucose is administered and a 50 min dynamic PET scan is started. After the scan, insulin infusion is discontinued and participants are monitored until plasma glucose levels are adequate for safe discharge.

For a subgroup of participants, skeletal muscle microvascular bloodflow will also be assessed with contrast-enhanced ultrasound performed during fasting and 30 minutes after the start of clamp. The participants will be administered intravenous contrast agent, and after steady plasma concentration is reached (2.5 min), the contrast agent micro bubbles are destroyed with a high-intensity ultrasound signal, and the rate at which small arterioles are refilled is measured.

Data will be analysed using in-house developed programs. Regions of interest will be drawn manually for peripheral tissues (skeletal muscle, visceral, brown and subcutaneous adipose tissue, liver, kidney, intestines) and using automated segmentation tools for the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-60 years
2. BMI either 18.5-25 kg/m2 or above 30 kg/m2
3. Use of hormonal contraception for women in child bearing age

Exclusion Criteria:

1. In the lean group history of obesity or type 2 diabetes
2. In the group with obesity: current or previous use of GLP-1-agonists or insulin
3. History of eating disorders
4. Smoking, use of narcotics, excessive use of alcohol
5. Previous participation in PET studies
6. Previous significant exposure to radiation
7. Claustrophobia
8. Active plans for concieving (both sexes)
9. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Insulin-induced change in tissue blood flow | Change from fasting condition to 10 minutes and 50 minutes after the start of insulin infusion
  Brain, liver, skeletal muscle and brain blood-flow (ml/100 g/min) measured with H2[15O]O PET/CT

SECONDARY OUTCOMES:
Effects of insulin on skeletal muscle microvascular perfusion | Change from fasting condition to 10 minutes and 50 minutes after the start of insulin infusion
  The difference in the rate of refill of skeletal muscle small capillaries measured as contrast agent wash-in using contrast-enhanced ultrasound during fasting and during hyperinsulinemic, euglycemic clamp
Tissue insulin-stimulated glucose uptake | Measured from 60 to 110 minutes after the start of insulin infusion
  Skeletal muscle, adipose tissue, liver and brain glucose uptake (micromol/100g/min) during hyperinsulinemic, euglycemic clamp measured with [18F]FDG PET/CT
Effects of emotions on whole-body blood flow | Measured during 60-second activation blocks (visual stimuli) or during 5 min cold-exposure
  Distribution of whole-body blood flow after visual stimuluses or cold exposure
Range of effective and feasible radiowater doses with whole-body PET/CT | During repetitive H2[15O]O scans (a total of 120 minutes)
  Repeatability and reliability of different doses of H2[15O]O in assessing tissue blood flow in the brain, skeletal muscle, myocardium, liver and adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Nummenmaa, Professor, Principal Investigator — University of Turku; Pirjo Nuutila, professor, Principal Investigator — University of Turku, Turku University Hospital
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT06739473/Prot_SAP_000.pdf